CLINICAL TRIAL: NCT01495390
Title: A Multicenter Study for the Discovery and Validation of ALS Biomarkers
Brief Title: A Longitudinal Study of Amyotrophic Lateral Sclerosis (ALS) Biomarkers
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Association (Other); ALS Finding a Cure (Other)
Responsible Party: Principal Investigator, James D. Berry MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: BIO-ALS-02
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Nervous System Diseases; Sclerosis; Motor Neuron Disease; Spinal Cord Diseases; Central Nervous System Diseases; Neurodegenerative Diseases; Neuromuscular Diseases; ALS
Keywords: Biomarkers; Biological Markers; Surrogate Markers; Clinical Markers; Plasma; Cerebrospinal Fluid; DNA; Serum; RNA
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Nervous System Diseases; Sclerosis; Motor Neuron Disease; Spinal Cord Diseases; Central Nervous System Diseases; Neurodegenerative Diseases; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples will be collected from participants with ALS over time. These biological samples include blood (plasma, serum, and RNA) and cerebrospinal fluid (CSF). DNA will be collected at one time point.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to collect biofluid samples for the banking and usage in ALS research. Through comparison of these samples, the researchers hope to learn more about the underlying cause of ALS, as well as find unique biological markers, which could be used to develop new therapies.

DETAILED DESCRIPTION:
The purpose of the research study is to collect blood samples and cerebrospinal fluid (CSF) from people with amyotrophic lateral sclerosis (ALS). These samples will be collected approximately every 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of suspected, possible, probable or definite ALS according to El Escorial Criteria
* Vital capacity (VC) at least 50 percent predicted
* Able to undergo multiple lumbar punctures

Exclusion Criteria:

* Abnormal CSF pressure or intracranial/intraspinal tumors
* Use of anticoagulant medication that cannot be safely withheld
* Bleeding disorders

  * This is a partial listing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers will be invited to participate in this study by their neurologists either in clinic or at a regular scheduled appointment visit
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2011-11; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale | Approximately every 4 months
  The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
Vital Capacity (VC) | Approximately every 4 months
  The vital capacity (VC) (percent of predicted normal) was determined using the slow VC method. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as a percent of predicted normal.
Hand Held Dynamometry (HHD) | Approximately every 4 months
  Hand Held Dynamometry (HHD) will be used as a quantitative measure of muscle strength for this study. Six proximal muscle groups will be examined bilaterally in both upper and lower extremities (shoulder flexion, elbow flexion, elbow extension, hip flexion, knee flexion, and knee extension), all of which have been validated against maximum voluntary isometric contraction (MVIC) testing.
Ashworth Spasticity Scale | Approximately every 4 months
  This is a standard measure for spasticity, has been used in a previous ALS clinical trials, and is applied in the current trial to evaluate the progression of spasticity due to upper motor neuron dysfunction in ALS.
Fronto-Temporal Dementia (FTD) Assessment | Approximately every 4 months
  The FTD Screening Assessment is a quickly administered scale used to evaluate memory, executive functions, and language. It is aimed at determining the presence of subtle dysfunction of these domains of cognition and behavior that may portend the onset of FTD or FTD-like symptoms.
ALS Cognitive Behavioral Screen (ALS CBS) | Approximately every 4 months
  The ALS Cognitive Behavioral Screen (ALS-CBS™) is a short measure of cognition and behavior in patients with Amyotrophic Lateral Sclerosis (ALS). The cognitive section includes commonly used elements of standard testing batteries, consisting of 8 tasks, with a possible total score of 20. It can be administered by a physician or other clinical care staff and takes approximately 5 minutes to complete.
  The behavioral section (ALS Caregiver Behavioral Questionnaire) is composed of questions sensitive to organic brain changes. It consists of a set of questions that compare changes in personality and behavior since the onset of ALS, as well as yes/no questions about mood, pseudobulbar affect, and fatigue. It is completed by a caregiver, family member or other informant during the same time that the patient completes the cognitive portion. The questionnaire typically takes about 2 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: James D. Berry, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Northeast ALS Consortium Website — http://www.alsconsortium.org